CLINICAL TRIAL: NCT02404935
Title: Randomized Phase II Study of First-line FOLFIRI Plus Cetuximab for 8 Cycles Followed by Either Single-agent Cetuximab as Maintenance Therapy or Observation in Patients With Wild-type KRAS and NRAS Metastatic Colorectal Cancer
Brief Title: Treatment After Irinotecan-based Frontline Therapy: Maintenance With Erbitux (in Patients wtRAS mCRC)
Acronym: TIME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prodige 28 - UCGI 27 (TIME); 2012-005139-99 (EudraCT Number)
Record Dates: First submitted 2015-03-23; First posted 2015-04-01 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; cetuximab; maintenance
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A cetuximab (Experimental): cetuximab 500 mg/m2 (every 2 weeks) until progression
  Interventions: Drug: Cetuximab; Drug: FOLFIRI and cetuximab
- Arm B observation (Other): observation until progression
  Interventions: Drug: FOLFIRI and cetuximab

INTERVENTIONS:
Drug: Cetuximab
  Arms: Arm A cetuximab
Drug: FOLFIRI and cetuximab

SUMMARY:
National multicentric phase II trial evaluating whether single agent cetuximab is effective as maintenance therapy after 8 cycles of first line FOLFIRI plus cetuximab in mCRC patients with KRAS and NRAS wild-type genes, assessed by progression-free survival at 6 months after start of maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal cancer
2. KRAS and NRAS wild-type genes after analysis of mutation status from the primary tumour or metastasis
3. Non resectable metastatic disease in a curative intent
4. No prior chemotherapy except for fluoropyrimidines with or without oxaliplatin-based adjuvant treatment, at least 6 months before inclusion
5. At least one measurable tumour target (higher than 20 mm) according to RECIST criteria, which has never been irradiated
6. Life expectancy above 3 months
7. Performance Status ≤2 (WHO)
8. Patient ≥18 years-old
9. Acceptable blood test
10. Patient having signed a written informed consent form

Exclusion Criteria:

1. Known and/or symptomatic brain metastases
2. Known allergy to one of treatment components
3. Neurological or psychiatric condition which could interfere with good treatment compliance
4. Current anti-tumour treatment : chemotherapy or targeted therapy or radiotherapy ≤ 14 days before randomisation
5. Other severe conditions such as: respiratory failure. History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan
6. Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) 6 months before enrollment/randomization
7. Concomitant severe infection
8. History of cancer (except skin cancer other than melanoma or an in situ cervical epithelioma or other solid tumour treated for curative purposes without signs of the condition and with no treatment administered in the 5 years before randomisation.)
9. Patient already included in another clinical trial with an investigational molecule
10. Prior treatment with anti-EGFr antibodies (e.g. panitumumab (Vectibix® or cetuximab / Erbitux® ) or treatment with small EGFr inhibitor molecules (e.g., erlotinib / Tarceva®)
11. Pregnant female, likely to be or currently breastfeeding, or planning to become pregnant within 6 months after the end of treatment or absence of effective contraception for males and females of childbearing age during treatment and for 6 months (male or female) after the end of treatment
12. Those deprived of their freedom or under guardianship
13. Impossibility of undergoing trial's medical follow-up for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2013-11-22 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival at 6 months | 6 months after start of maintenance therapy
  Endpoints will include Progression assessed by CT Scan according to RECIST 1.1 criteria and Death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Boige, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (46):
- France (46):
  - CHU- Hôpital Sud, Amiens
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier d'Auxerre, Auxerre
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier Intercommunal Cote Basque, Bayonne
  - Centre Hospitalier de Beauvais, Beauvais
  - Centre Hospitalier de Béziers, Béziers
  - Centre Hospitalier de Blois, Blois
  - Hôpital Avicenne, Bobigny
  - Clinqiue Tivoli, Bordeaux
  - Institut Bergonie, Bordeaux
  - Centre François Baclesse, Caen
  - Hôpital Côte de nacre, Caen
  - Centre Hospitalier Jean Rougier, Cahors
  - Centre Hospitalier Estaing, Clermont-Ferrand
  - Hôpital du Bocage, Dijon
  - Centre Hospitalier de la Dracénie, Draguignan
  - Clinique du Mousseau, Évry
  - Centre Hospitalier Intercommunal, Fréjus
  - Centre hospitalier Départemental de Vendée - Les Oudairies, La Roche-sur-Yon
  - Clinique du Cap d'Or, La Seyne-sur-Mer
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Centre Oscar Lambret, Lille
  - Clinique Francois Chenieux, Limoges
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Clairval, Marseille
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier Montelimar, Montélimar
  - Centre de Cancérologie du Grand Montpellier - Clinique Clementville, Montpellier
  - Institut régional du Cancer Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier d'Orléans La Source, Orléans
  - Hôpital Saint Jean, Perpignan
  - Polyclinique Francheville, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU - Robert Debre, Reims
  - Centre Hospitalier de Romans, Romans
  - Centre Hospitalier Hôpital Victor Provo, Roubaix
  - Hôpital Saint Gregoire, Saint-Grégoire
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - CHU Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Polyclinique de l'Ormeau, Tarbes
  - Centre Hospitalier Intercommunal de Toulon, Toulon
  - Gustave Roussy, Villejuif, Île-de-France Region

REFERENCES:
- [Derived] Boige V, Blons H, Francois E, Ben Abdelghani M, Phelip JM, Le Brun-Ly V, Mineur L, Galais MP, Villing AL, Hautefeuille V, Miglianico L, De La Fouchardiere C, Genet D, Levasseur N, Levache CB, Penel N, Mitry E, Jacquot S, Aparicio T, Brument E, Gourgou S, Castan F, Bouche O. Maintenance Therapy With Cetuximab After FOLFIRI Plus Cetuximab for RAS Wild-Type Metastatic Colorectal Cancer: A Phase 2 Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2333533. doi: 10.1001/jamanetworkopen.2023.33533. PMID 37721754